CLINICAL TRIAL: NCT06202846
Title: Identification of Y Chromosome From Free Circulating DNA in Patients With Turner Syndrome
Acronym: Turner-Ylc
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 8788
Record Dates: First submitted 2023-10-20; First posted 2024-01-12 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Turner Syndrome
Keywords: Turner syndrome; Y chromosome
MeSH Terms: conditions — Turner Syndrome

STUDY DESIGN:
Intervention Model Description: * Plasma isolated from whole blood sampled on BCT strecl tube
  * Whole blood sampled on heparin tube
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Turner syndrome patients (Experimental): Patients with a Turner syndrome confirmed by karyotype.
  Interventions: Genetic: cfDNA analysis

INTERVENTIONS:
Genetic: cfDNA analysis — In order to compare the performance of the ctDNA test with techniques used in routine diagnostics, we will compare the results obtained by the ctDNA test with those obtained by FISH.
  compare the results obtained by the ctDNA test and FISH. This will enable us to identify a potential diagnostic gain. We will compare the percentage of patients for whom a positive test result result was obtained by the lncDNA test (Y chromosome detection) to the percentage of patients for whom a positive result was obtained by FISH.

SUMMARY:
Turner syndrome affects 1/2500 female newborns. It is characterized by a short stature, gonadal dysgenesis and bone anomalies. It is secondary to X chromosome abnormality. The clinical course can be marked by various complications, including degeneration of gonadal streaks into cancer (gonadoblastoma). The risk of gonadoblastoma is increased by the presence of Y chromosome, with a risk of 19 to 43%. However, Y chromosome material may be difficult to identify due to its mosaic state, at varying rates depending on the tissue. Free circulating DNA (cfDNA) corresponds to fragments of extracellular DNA present in the plasma, released into the circulation during cell death processes by the various tissues of the body. Due to its multiple tissue origins and easy collection, cfDNA appears to be a suitable matrix for searching for low mosaic Y chromosome sequences in patients with Turner syndrome.

The main objective of the study is to develop a cfDNA-based test to look for Y chromosome sequences in 50 patients with Turner syndrome. The secondary objectives are to determine the mosaic detection threshold of this test and to compare the performance of this test with the fluorescence in situ hybridization (FISH) technique used in routine diagnosis.

This study will assess the detection sensitivity of this test and its relevance in a clinical context.

ELIGIBILITY:
Inclusion Criteria:

* patient aged 2 to 74 years
* with a diagnosis of Turner syndrome confirmed by karyotype
* who have given their consent or whose legal representative(s) have given their consent(s) consent(s) to participate in the study
* affiliated to the French Social Security system or benefiting from such a system

Exclusion Criteria:

* male phenotype
* patient or legal representative(s) with comprehension difficulties (linguistic, etc.)
* patients covered by articles L.1121-5 to L.1121-8 of the CSP (French Public Health Code)

Ages: 2 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients presenting Y chromosome material detected by the cfDNA test | From date of inclusion to date of genetic analysis result
  An inferential analysis will allow to estimate the proportion of Y chromosome detection by the cfDNA test and secondly to compare it with data from the literature.

SECONDARY OUTCOMES:
Y chromosome mosaic rate detectable by the cfDNA test. | Up to 26 months
  Dilution of female (XX) and male (XY) plasma in order to evaluate the detection limit of y chromosome material by the cfDNA test.
Comparison between the cfDNA test and routine FISH analysis | Up to 30 months
  An inferential analysis will compare the proportion of Y chromosome detection by the cfDNA test and by FISH.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hospice Civil de Lyon, Lyon
  - Hopitaux Universitaire de strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No